CLINICAL TRIAL: NCT07385261
Title: Treatment Strategy for Complicated Pediatric Appendicitis Based on Laparoscopic Surgery. Ten Years of Multicenter Cohort Study
Brief Title: Treatment Strategy for Complicated Pediatric Appendicitis Based on Laparoscopic Surgery
Acronym: CALAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Daboos (Other)
Collaborators: South Valley University (Other); Tanta University (Other)
Responsible Party: Sponsor-Investigator, Mohammad Daboos, Assistant professor of pediatric surgery, Faculty of Medicine, Al-Azhar University, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUV-MED- SUR011-4-25-3-2
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Appendix Diseases; Surgery
Keywords: laparoscopic surgery; complicated appendicitis

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Pediatric patients aged less than 18 years, with Complicated appendicitis (with mass, appendicular abscess, and free collection) received surgical intervention with laparoscopy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complicated Appendicitis (Experimental): Complicated appendicitis: refer to acute appendicitis with perforation or gangrene, appendicular mass with or without abdominal abscess formation submitted for laparoscopic management with appendectomy and intraperitoneal suction of pus over the last 10 years
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Procedure: laparoscopic appendectomy — Based on clinical findings, imaging studies and laboratory findings, after resuscitation, the decision of urgent surgery was according to the presentation Free peritoneal perforation (FPA) Perforated appendicitis with free peritoneal fluid were managed by urgent laparoscopic exploration Appendicular mass (AM) In patients presented by early mass formation lap exploration was carried out but trial of conservative management was planned for cases presented late with expected difficulty in lap dissection depending on surgical team and parental consultation, this accomplished by (nothing per mouth, I V fluid, I V antibiotic, temperature chart with U/S and biomarker follow up)
  Appendicular abscess (AAbs) Percutaneous drainage by availability IR team was the first choice however lap exploration and /or lap assisted extraperitoneal drainage was the second choice if IR failed or not available.

SUMMARY:
Observational retrospective study included 765 children with Operative management by laparoscopic appendectomy, conservative management for appendicular mass and drainage of abscess by IR should be tried first. Interval appendectomy is reserved only for patients with recurrent symptoms. the study collect the Diagnostic data ,intraoperative and post operative data to submit the strategies of laparoscopic management in limited resources setting.

DETAILED DESCRIPTION:
Background and study aims: In children with complicated appendicitis significant morbidity exists with prolonged hospitalization and increased costs. The management strategy for complicated pediatric appendicitis differs depending on facility resources together with surgeon's experience. Various studies investigated the usefulness of laparoscopic than open surgery even in complicated appendicitis. However, the treatment strategy remains controversial, especially in appendicular mass as well as appendicular abscess.

Methods: This observational study included 765 children with complicated appendicitis. over 10 years period. Patients' demographics, clinical criteria for different presentations of complicated appendicitis, diagnostic work up, plans of treatment based on laparoscopic management were reviewed and analyzed regarding different variables and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic management of Complicated Appendicitis with mass formation
* laparoscopic management of Complicated appendicitis with abscess formation:
* laparoscopic management of Complicated appendicitis with free intraperitoneal collection

Exclusion Criteria:

* Open surgery cases
* Patients received incomplete antibiotic therapy
* Accidental discovery coexistent pathology that necessitates open surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 765 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Primary outcomes | 4 years
  postoperative outcomes any alarming symptoms of intestinal obstruction developed (vomiting, fever, or severe abdominal pain, intraperitoneal collections

CONTACTS AND LOCATIONS:
Overall Officials: ‪Mohammad Daboos‬, Dr, Principal Investigator — Department of pediatric surgery, faculty of medicine , Al-Azhar University
Locations (1):
- Mohammad Daboos, Cairo, Egypt